CLINICAL TRIAL: NCT00168363
Title: Safety and Efficacy of Brimonidine in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-022
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate

INTERVENTIONS:
Drug: brimonidine

SUMMARY:
This Study will evaluate the safety and efficacy of brimonidine in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* ocular hypertension or glaucoma in both eyes
* currently treated with brimonidine
* requires IOP-lowering therapy in both eyes

Exclusion Criteria:

* uncontrolled systemic disease
* known allergy or sensitivity to brimonidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
lowering of intraocular pressure

REFERENCES:
- [Derived] Cantor LB, Safyan E, Liu CC, Batoosingh AL. Brimonidine-purite 0.1% versus brimonidine-purite 0.15% twice daily in glaucoma or ocular hypertension: a 12-month randomized trial. Curr Med Res Opin. 2008 Jul;24(7):2035-43. doi: 10.1185/03007990802199287. Epub 2008 Jun 4. PMID 18534052
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com